CLINICAL TRIAL: NCT01315379
Title: Prolonged Exposure Therapy (PE) for Post-traumatic Stress Symptoms and Mild TBI Symptoms in Children Following Motor Vehicle Accident.
Brief Title: Psychological Treatment for Children Suffering From Post Traumatic Stress Symptoms and Mild Traumatic Brain Injury
Acronym: TBI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 6166
Record Dates: First submitted 2011-03-03; First posted 2011-03-15 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: PTSD; Traumatic Brain Injury; Post Concussive Syndrome
Keywords: Prolonged Exposure; CBT; PTSD; Mild Traumatic Brain Injury; Post Concussive Syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Post-Concussion Syndrome; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PTSD without TBI: children and adolescents with a diagnosis of PTSD and without head injury, following a motor vehicle accident.
  This group will be treated using the Prolonged Exposure Therapy protocol.
  Interventions: Behavioral: Prolonged Exposure Therapy
- PTSD with m-TBI: children and adolescents with a diagnosis of PTSD and a diagnosis of mild traumatic brain injury, following a motor vehicle accident.
  This group will be treated using the Prolonged Exposure Therapy protocol.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — This intervention comprises 12-18 sessions of cognitive behavior therapy for PTSD with the components (a) Psychological education, (b) in vivo exposure (c) prolonged imaginal exposure, (d) cognitive restructuring (e) summary and relapse prevention.

SUMMARY:
The purpose of this study is to determine whether Prolonged Exposure Therapy (PE)is effective in the treatment of post-traumatic stress symptoms in children and adolescents with mild traumatic brain injury (m-TBI) due to motor vehicle accident.

DETAILED DESCRIPTION:
Motor vehicle accidents account for a majority of TBI cases and are a leading cause for Post Traumatic Stress Disorder (PTSD) among children. The vast majority of these cases involve mild TBI (mTBI) with persistent post concussion syndromes. However, the empirical data on treatment in this field is scarce. Few studies demonstrated that cognitive behavioral therapies can be effective for adults with mild TBI suffering from Acute Stress Disorder, but no research, to date, addressed this question in pediatric population. In the current research we intend to examine the effectiveness of PE in reducing post-traumatic stress symptoms in children and adolescents with m-TBI caused by motor vehicle accident, in comparison to children and adolescents without brain injury.

Sixty children age 6 to 18 attending the Anxiety clinic in Schneider Children's Medical Center of Israel will be included. All subjects will be treated with a manualized 12-18 week Prolonged Exposure protocol. Participants will undergo assessments, which will include interviews, questionnaires and neuropsychological tests concerning symptoms of PTSD, emotional and cognitive functioning. Ratings and neuropsychological testing will be made at baseline and following completion of treatment. Follow up will include questionnaires ratings at 2 weeks, 4 weeks and 12 weeks after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

For the whole sample:

* Children age 6 to 18
* Language spoken: Hebrew, Arabic
* DSM- IV R diagnosis: PTSD
* Car accident event within past 3 years

For the m-TBI group:

* Any of the following symptoms or experiences occurring during or shortly after the accident: loss of consciousness, dazed, confused, saw stars, headache, dizziness, irritability, memory gap (not remembering injury or injury period), visual loss, abdominal pain].
* Diagnosis of MTBI within 3 years as confirmed by CT/MRI/fMRI.
* Glasgow coma scale; GCS<15.

Exclusion Criteria:

* Children presenting with psychotic symptoms
* Children presenting with mental retardation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sixty children age 6 to 18 attending the Anxiety clinic in Schneider Children's Medical Center of Israel, following MVA, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with PTSD diagnosis as a measure of recovery rates | After up to 18 weeks of PE treatment
  Psychological evaluation using the Hebrew translation of the Childhood version of the Schedule for Affective Disorders and Schizophrenia (Apter et al., 1989).

SECONDARY OUTCOMES:
Change from Baseline in Neuropsychological Functioning at Treatment Completion | After up to 18 weeks of treatment
  Subjects will take paper and pencil and computer tests to evaluate memory, learning, attention and concentration, vocabulary and naming.
  The neuropsychological testing battery includes: Raven's Progressive Matrices, BRIEF, WISC-III-Hebrew Version (Digit Span), CMS (Spatial Span), D-KEFS (Design Fluency, Sorting Test, Trails Making Test), CPT, Stroop,TOMM Effort validity test, The Connors Rating Scale- Revised Long version
Change from Baseline in The Child PTSD Symptoms Scale at Treatment Completion | At up to 18 weeks of PE treatment
  The Child PTSD Symptoms Scale (Foa et al., 2001)
Change from Baseline in The Child PTSD Symptoms Scale at 2 weeks Follow Up | 2 weeks following treatment completion
  The Child PTSD Symptoms Scale (Foa et al., 2001)
Change from Baseline in The Child PTSD Symptoms Scale at 4 weeks Follow Up | 4 weeks following treatment Completion
  The Child PTSD Symptoms Scale (Foa et al., 2001)
Change from Baseline in The Child PTSD Symptoms Scale at 12 weeks Follow Up | 12 weeks following treatment completion
  The Child PTSD Symptoms Scale (Foa et al., 2001)
Change from Baseline in the Childrens Depression Inventory at Treatment Completion | After up to 18 weeks of PE treatment
  Childrens Depression Inventory, Kovacs, 1992
Change from Baseline in the Children's Global Assessment Scale at Treatment Completion | After up to 18 weeks of PE treatment
Change from Baseline in The State-Trait Anxiety Inventory for Children at Treatment Completion | After up to 18 weeks of PE Treatment
  The State-Trait Anxiety Inventory for Children, Spielberger et al.
Change from Baseline in The Well-Being Questionnaire at Treatment Completion | After up to 18 weeks of PE treatment
  WHO-5 (Bech, 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Maayans Shorer, PhD, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No